CLINICAL TRIAL: NCT01139905
Title: Pharmacokinetics of Low- Dose Lopinavir/Ritonavir Tablet Formulation HIV-1 Infected Children
Brief Title: Lopinavir/Ritonavir (LPV/r) Tablet in HIV Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HIV-NAT 100
Record Dates: First submitted 2010-06-04; First posted 2010-06-09 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: HIV-1 Infections
Keywords: Lopinavir/ritonavir; pharmacokinetic; low dose; HIV-infected children; pharmacokinetics of low-dose lopinavir/ritonavir in HIV-1 infected Thai children.
MeSH Terms: interventions — Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): standard dose of lopinavir/ritonavir 100/25 mg tablet q 12 hour
  Interventions: Other: lopinavir/ritonavir

INTERVENTIONS:
Other: lopinavir/ritonavir — standard dose of lopinavir/ritonavir 100/25 mg tablet q 12 hour.

SUMMARY:
To study the pharmacokinetics of low-dose lopinavir/ritonavir tablet in HIV-1 infected Thai children.

DETAILED DESCRIPTION:
This is an open-label, single arm study to compare standard dose with a new tablet formulation of a lower dose of lopinavir/ritonavir in HIV-1 infected children.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection
2. Age < 18 years old
3. BW > 25 kg
4. HIV RNA viral load < 50 copies within 6 months
5. Written informed consent

Exclusion Criteria:

1. Active opportunistic infection
2. Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.
3. Use of concomitant medications that may interfere with the pharmacokinetics of lopinavir/ritonavir

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
assess the level of lopinavir trough level >1 mg/L in low dose lopinavir (reduction by 70%) | 4 months
  study drug Aluvia (lopinavir/ritonavir 100/25 mg)

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT, Bangkok, Thailand

REFERENCES:
- [Result] Klinklom A, Puthanakit T, Gorowara M, Phasomsap C, Kerr S, Sriheara C, Ananworanich J, Burger D, Ruxrungtham K, Pancharoen C. Low dose lopinavir/ritonavir tablet achieves adequate pharmacokinetic parameters in HIV-infected Thai adolescents. Antivir Ther. 2012;17(2):283-9. doi: 10.3851/IMP1958. Epub 2011 Nov 10. PMID 22293065
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org